CLINICAL TRIAL: NCT05217966
Title: Single Pre-Operative Radiation Therapy - With Delayed or No Surgery (SPORT-DNS) for Low Risk Breast Cancer: A Phase II Study
Brief Title: Single Pre-Operative Radiation Therapy - With Delayed or No Surgery (SPORT-DNS)
Acronym: SPORT-DNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Michael Yassa, Radiation Oncologist, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-12-2021-2565
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: ablative radiotherapy; preoperative radiotherapy; neoadjuvant radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative radiotherapy for early breast cancer (Experimental): Radiation: Single Pre-Operative Radiation Therapy
  Interventions: Radiation: Radiation: Single Pre-Operative Radiation Therapy

INTERVENTIONS:
Radiation: Radiation: Single Pre-Operative Radiation Therapy — Ablative preoperative partial breast radiation therapy

SUMMARY:
Eligible women will receive neoadjuvant single fraction radiotherapy followed by surgery performed after one year

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 50 years or older.
2. Postmenopausal status (Defined as: age 60 OR bilateral ovariectomy OR amenorrhea > 12 months prior to breast cancer diagnosis without using oral contraceptives/hormone replacement therapy) (65).
3. World Health Organization (WHO) performance status 0-2.
4. Invasive ductal carcinoma proven by biopsy done ≤ 12 weeks from treatment start.
5. Unifocal disease on preoperative staging ultrasound or MRI done ≤ 12 weeks from treatment start.
6. Tumors less than or equal to 2cm clinically on physical exam, as well as on breast ultrasound.
7. No clinical evidence of nodal disease (i.e. cN0), on physical examination done ≤ 12 weeks from treatment start, as well as on breast ultrasound.
8. Estrogen receptor status (ER) positive on biopsy ≥ 80%.
9. Progesterone receptor status (PR) positive on biopsy ≥ 20%.
10. Her2 negative on biopsy.
11. No lymphovascular invasion on biopsy.
12. Low Oncotype DX recurrence score performed on biopsy specimen (RS ≤18).
13. Planned surgery is a partial mastectomy with sentinel lymph node biopsy.

Exclusion Criteria:

1. Age less than 50 years.
2. Premenopausal or uncertain menopausal status.
3. A known deleterious mutation in BRCA 1 and/or BRCA 2.
4. Clinical tumor size > 2.0 cm in greatest diameter on staging ultrasound.
5. Tumor histology limited to lobular carcinoma only.
6. Clinically positive axillary nodes (cN+).
7. Lymphovascular invasion on biopsy.
8. Pure ductal or lobular carcinoma in situ on biopsy.
9. Extensive intraductal component on biopsy.
10. Neoadjuvant hormonal manipulation or chemotherapy.
11. Prior non basal cell or squamous cell skin cancers within 5 years.
12. More than one primary tumor in different quadrants of the same breast.
13. Diffuse microcalcifications on mammography.
14. Paget's disease of the nipple.
15. Previous irradiation to the ipsilateral breast.
16. Presence of an ipsilateral breast implant or pacemaker.
17. Serious non-malignant disease (e.g. cardiovascular, pulmonary, systemic lupus erythematosus (SLE), scleroderma) which would preclude definitive radiation treatment.
18. Estrogen receptor status (ER) not known.
19. Currently pregnant or lactating.
20. Psychiatric or addictive disorders which would preclude obtaining informed consent or adherence to protocol.
21. Geographic inaccessibility for follow-up.
22. Lack of preoperative staging with breast and axillary ultrasound.
23. Inability to adequately plan the patient for the experimental technique.
24. Prior breast cancer.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pathological complete response | 12 months

SECONDARY OUTCOMES:
Incidence of grade 3 or greater radiation toxicity | 0-5 years

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided